CLINICAL TRIAL: NCT04220723
Title: Evaluation of Frailty and Functional Capacity in End-Stage Liver Disease
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Bilge Taskin Gurel, Msc PT, Hacettepe University
Other Study IDs: ESLD
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: End Stage Liver Disease
Keywords: end stage liver disease; frailty; exercise test; muscle weakness; exercise tolerance; hand strength; muscle strength
MeSH Terms: conditions — End Stage Liver Disease; Frailty; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- End-Stage Liver Disease: End-stage liver disease patients who are being followed up at the Department of Gastroentereology of Hacettepe University Faculty of Medicine will be included in the study. When the participants come to the gastroenterology department for control, they will be directed to us and the assessment will begin after written and verbal approval is obtained. The Liver Frailty Index will be used to assess the frailty of the participants. Accordingly, hand grip test, 5 repeat sit-up test and side, semi-tandem and tandem balance measurements will be made and a total frailty score will be obtained. Submaximal aerobic capacities and functional capacities will be evaluated by 6 Minute Walk Test. Then, maximal inspiratory muscle pressure and maximal expiratory muscle pressure of the participants will be measured and respiratory muscle strength will be evaluated. Finally, maximal aerobic capacity will be measured by Shuttle Walk Test.
  Interventions: Other: Frailty Assessment; Other: Functional Capacity Assessment

INTERVENTIONS:
Other: Frailty Assessment — Liver Frailty Index measurements:
  1. Grip strength: the average of three trials, measured in the subject's dominant hand using a hand dynamometer
  2. Timed chair stands: measured as the number of seconds it takes to do five chair stands with the subject's arms folded across the chest
  3. Balance testing: measured as the number of seconds that the subject can balance in three positions (feet placed side-to-side, semitandem, and tandem) for a maximum of 10 seconds each.
Other: Functional Capacity Assessment — Shuttle Walk Test: The patient is required to walk around two cones set 9 metres apart (so the final track is 10 metres) in time to a set of auditory beeps played on a CD. Initially, the walking speed is very slow, but each minute the required walking speed progressively increases. The patient walks for as long as they can until they are either too breathless or can no longer keep up with the beeps, at which time the test ends. The number of shuttles is recorded. Each shuttle represents a distance of ten metres (i.e each time the patient reaches a cone is 1 shuttle).

SUMMARY:
Development of fibrosis plays a main role in the pathophysiology of liver diseases. The rate of progression in fibrogenesis varies according to the type of underlying liver disease and varies with the environment and host-related factors. End-stage liver diseases are characterized by systemic vascular resistance and decreased arterial blood pressure, increased heart rate and cardiac output . Disruption of regulation of neurogenic, humoral and vascular functions is effective in these cardiovascular changes. In end-stage liver diseases, glycogen storage and corruption of glyconeogenesis cause muscle protein and fat to be used for energy, resulting in weight loss and muscle weakness. According to the latest data of the Republic of Turkey Ministry of Health in Turkey in 2223 patients are waiting for liver transplantation. Acute and chronic liver disease and infectious complications lead to an increase in the number of hospitalizations and prolonged hospital stay and severely affect the functional status and mortality. In recent years, more attention has been paid to complications from chronic diseases, including malnutrition, sarcopenia, poor functional capacity, and frailty. There are few studies in the literature examining functional capacity and physical frailty in end-stage liver disease. The aim of this study was to investigate the relationship between functional capacity and frailty in end-stage liver disease.

DETAILED DESCRIPTION:
The decrease in functional capacity is a finding that affects quality of life in chronic liver diseases. In a study, 6 Minute Walk Test was associated with mortality in patients with cirrhosis and survival was lower in patients walking less than 250 meters. Malnutrition is a common complication of end-stage liver disease. It is a complex condition that causes loss of muscle and fat mass, loss of body weight, increased pro-inflammatory cytokines, anorexia and fatigue, resulting in sarcopenia. Sarcopenia is generally defined as a loss of muscle mass and muscle strength and is directly related to adverse outcomes in these patients. In the evaluation of malnutrition in end-stage liver disease, evaluation of skeletal muscle (mass, strength, functionality) provides an objective way to determine malnutrition, since most intrinsic markers originate from existing liver disease (eg albumin, prealbumin, lymphopenia levels).

ELIGIBILITY:
Inclusion Criteria:

* Follow-up with end-stage liver disease in Hacettepe University Faculty of Medicine, Department of Gastroenterology
* Volunteering for research

Exclusion Criteria:

* Presence of hepatopulmonary syndrome
* Presence of portopulmonary hypertension
* Uncontrolled severe hepatic encephalopathy
* Previous history of liver transplantation
* Presence of orthopedic problems that will affect the research
* Presence of neurological deficits
* Severe chronic obstructive pulmonary disease or heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population defined as decompanse or companse cirrhosis that caused end-stage liver disease.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Frailty | 10 minutes
  Liver Frailty Index used to assess frailty. Accordingly, hand grip test, 5 repeat sit-up test and side, semi-tandem and tandem balance measurements will be made and a total frailty score will be obtained.
Functional Capacity | 20 minutes
  Shuttle Walk Test used to assess maximal aerobic capacity. The patient is required to walk around two cones set 9 metres apart (so the final track is 10 metres) in time to a set of auditory beeps played on a CD. Initially, the walking speed is very slow, but each minute the required walking speed progressively increases. The patient walks for as long as they can until they are either too breathless or can no longer keep up with the beeps, at which time the test ends. The number of shuttles is recorded. Each shuttle represents a distance of ten metres.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Taşkın, MS PT, Principal Investigator — Hacettepe University Faculty of Physical Therapy and Rehabilitation; Naciye Vardar-Yağlı, PhD, Study Chair — Hacettepe University Faculty of Physical Therapy and Rehabilitation; Ahmet Bülent Doğrul, MD PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernal W, Martin-Mateos R, Lipcsey M, Tallis C, Woodsford K, McPhail MJ, Willars C, Auzinger G, Sizer E, Heneghan M, Cottam S, Heaton N, Wendon J. Aerobic capacity during cardiopulmonary exercise testing and survival with and without liver transplantation for patients with chronic liver disease. Liver Transpl. 2014 Jan;20(1):54-62. doi: 10.1002/lt.23766. Epub 2013 Nov 29. PMID 24136710
- [Background] Duarte-Rojo A, Ruiz-Margain A, Montano-Loza AJ, Macias-Rodriguez RU, Ferrando A, Kim WR. Exercise and physical activity for patients with end-stage liver disease: Improving functional status and sarcopenia while on the transplant waiting list. Liver Transpl. 2018 Jan;24(1):122-139. doi: 10.1002/lt.24958. PMID 29024353